CLINICAL TRIAL: NCT02042742
Title: Effects of Punicalagin and Hydroxytyrosol Mixture on Different Inflammatory Markers Related With Cardiovascular Disease: a Crossover Study in Healthy Middle-aged Volunteers
Brief Title: Punicalagin and Hydroxytyrosol Mixture on Different Inflammatory Markers
Acronym: PROBELTEII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PROBELTEII
Record Dates: First submitted 2013-12-27; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Cross-over studies; Antioxidants; Hydroxytyrosol; Punicalagin; Treatment outcome; Inflammatory markers; Endothelial function; Humans; Adults; volunteers
MeSH Terms: interventions — punicalagin; 3,4-dihydroxyphenylethanol; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant supplement (Experimental): Treatment consist of consuming 65g of punicalagin and 3,3g of hydroxytyrosol (plus 331,7g of maltodextrin) three times daily, during 8 weeks.
  Interventions: Dietary Supplement: punicalagin and hydroxytyrosol mixture
- Control supplement (Placebo Comparator): Treatment consist of consuming 400g of maltodextrin three times daily, during 8 weeks.
  Interventions: Dietary Supplement: Control supplement (maltodextrin)

INTERVENTIONS:
Dietary Supplement: punicalagin and hydroxytyrosol mixture — Antioxidant Supplement (punicalagin and hydroxytyrosol mixture) During one period of crossover study (I or II) volunteers consume daily of functional supplement during 8 weeks. Additionally, volunteers must follow guidelines for healthy diet and physical activity.
  Other Names: Punicalagin and hydroxytyrosol
  Arms: Antioxidant supplement
Dietary Supplement: Control supplement (maltodextrin) — During one period of crossover study (I or II) volunteers consume daily of functional supplement during 8 weeks. Additionally, volunteers must follow guidelines for healthy diet and physical activity.
  Other Names: Maltodextrin
  Arms: Control supplement

SUMMARY:
A crossover trial was carried out in healthy volunteers aged 45-70 years and BMI <30 kg/m2. Subjects consumed a Antioxidant Supplement (AS) containing 65 mg of punicalagin mixed with 3.3 mg of hydroxytyrosol 3 times daily or a Control Supplement (CS) with maltodextrin for an 8 wk each phase with 4-wk rest period. Supplementation order was randomly assigned and the consumption of derivative products of punicalagin and/or hydroxytyrosol restricted. The endothelial function parameters (brachial artery flow-mediated dilation (FMD), biochemical markers), inflammatory markers and nutritional status were evaluated before and after each phase. Previously a pilot study was completed with no placebo (n=30) to determinate the effective dose of Functional Supplement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 45 to 75 years old;
* Signed informed consent

Exclusion Criteria:

* Individuals with cardiovascular risk factors on drug treatment (dyslipidemia, hypertension, Diabetes Mellitus);
* Individuals with Metabolic Syndrome;
* Individuals with familiar background of premature cardiovascular disease;
* Individuals with BMI ≥ 30 kg/m2;
* Women that still maintain your menstrual cycle;
* Individuals with increased alcohol consumption 30g/day;
* Individuals that stop smoking in the next 20 weeks (during the study);
* Individuals that consume antioxidant supplement, drugs, ω-3 supplements, vitamins, minerals, prebiotics or/and probiotics;
* Women that consume oral contraceptive;
* Individuals with mental disease or low cognitive function;
* Individuals with severe diseases (hepatic, kidney, cancer…);
* Individuals with drugs or supplements consumption to weight lost;
* Pregnant women or lactating;
* Individuals with intensive physical activity;
* Individuals with physical problems complying with the recommendations of physical activity and diet general recommendations.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in the Inflammatory markers after 8 weeks treatment | 0, 8, 12 and 20 weeks
  Inflammatory markers (Fibrinogen, gelsolin, thrombospondin, interleukin 6 and PCR) will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II

SECONDARY OUTCOMES:
Change in Oxidative Stress Parameters | 0, 8, 12 and 20 weeks
  Parameters measured were: plasma antioxidant capacity (FRAP, ferric reducing antioxidant power) and lipidic peroxidation (TBARS, thiobarbituric acid reactive substances assay), oxidized LDL, paraoxonase 1, F2-isoprostanes. Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II.
Change in Glucose Metabolism | 0, 8, 12 and 20 weeks
  Parameters measured were: glucose, basal insulin, HbA1c (in diabetic patients), HOMA (homeostasis model assessment ) index (glycemic insulin sensitivity index was calculated using the formula: HOMA-IR ( (homeostasis model assessment insulin resistance) = fasting glucose (mmol/l)/fasting immunoreactive insulin (mU/ml)/22•5).Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II
Change in Lipid profile | 0, 8, 12 and 20 weeks
  Parameters measured were: Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides. Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II
Change in Endothelial function | 0, 8, 12 and 20 weeks
  Parameters measured were: Brachial artery flow-mediated dilation (FMD), blood pressure, eNOS, vascular endothelial cell adhesion molecule -1 and p-selectin. Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II
Change in Coagulation markers | 0, 8, 12 and 20 weeks
  Parameters measured were: Prothrombin time and activity, INR. Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II
Change in Anthropometric and body composition parameters | 0, 8, 12 and 20 weeks
  Parameters measured were: Weight, Height and waist circumference, muscle mass percentage (MM%), fat mass percentage (FM%), free fat mass percentage(FM%). Will be measured at week 0 and 8 for phase I, and at week 12 and 20 for phase II
Adverse effects | 0 to 20 weeks
  Parameters measured were: transaminases and creatinine. Will be evaluated during all the study visits
Adherence and Tolerance Parameters | 0 to 20 weeks
  Parameters measured were: adherence and tolerance to the products. Will be evaluated during all study visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- See also: Institute for Health Research IdiPAZ — http://www.idipaz.es